CLINICAL TRIAL: NCT03205332
Title: An Experimental Investigation of the Effects of Concrete Thinking on Worry, Problem-Solving and Cognitive Processing in Individuals With Generalized Anxiety Disorder
Brief Title: Training Mental Habits Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Naomi Koerner, Associate Professor, Toronto Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-146-1
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2019-12

CONDITIONS: Generalized Anxiety; Worry
Keywords: Worry; Anxiety
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders

STUDY DESIGN:
Masking Description: Eligibility Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concreteness Training (Experimental): Participants receive 1 session of training in concrete processing during the pre-intervention visit. They are then asked to engage in 30 minutes of concreteness practice daily, for 7 days.
  Interventions: Behavioral: Concreteness Training
- Control (No Intervention): Assessment only.

INTERVENTIONS:
Behavioral: Concreteness Training
  Arms: Concreteness Training

SUMMARY:
Generalized Anxiety Disorder (GAD) is a chronic condition whose hallmark feature is excessive and uncontrollable worry (American Psychiatric Association, 2013). Theories of GAD propose that specific cognitive biases are involved in the maintenance and etiology of chronic worry. One cognitive bias that plays a role in worrying is abstract thinking, or the tendency to "verbalize" thoughts and worries in a manner that is vague and lacking in detail. There is evidence that training depressed people to think more concretely improves depressive symptoms and depression-type thinking styles, and reduces emotional reactivity. Given that chronic worry and depression have commonalities (e.g., repetitive thinking styles, difficulties with problem-solving and attentional control, emotion dysregulation), concreteness training may help people who struggle with chronic worry. The main goals of this proof of concept experiment are 1) to test in individuals reporting chronic worry the effects of an active form of concreteness training that involves imagery practice (compared to a no training control condition) on frequency of worrying, problem solving quality, and worry-related processes; 2) to examine the degree to which concreteness training causes improvements in daily worry and negative affect during the 7 days of practice. The study design will provide us with an understanding on a more "macro" level of the potential short-term benefits and will at the same time allow us to see, on a more "micro" level, how training concreteness affects worry and mood on a day-to-day basis during a 7-day period. The findings from this study will inform relevant clinical literature about efficacious methods to reduce chronic worry.

DETAILED DESCRIPTION:
The main goals of this proof of concept experiment are 1) to test in individuals reporting chronic worry the effects of an active form of concreteness training that involves imagery practice (compared to a no training control condition) on frequency of worrying, problem solving quality, and worry-related processes; 2) to examine the degree to which concreteness training causes improvements in daily worry and negative affect during the 7 days of practice. Participants are recruited from the community via advertisements. Following a telephone screen, participants attend a baseline visit during which they complete the MINI interview. Those who continue to be eligible complete the outcome measures and are randomly assigned to either the experimental condition or the control condition. Participants assigned to the experimental condition receive training in concrete processing and learn how to complete the daily experience sampling diary. Participants assigned to the control condition do not receive training and learn how to complete the daily experience sampling diary. All participants then complete their assigned activities for 7 days. They then return to the lab to complete the outcome measures at post-test, 1 week follow up and 1 month follow up. Participants are then debriefed.

ELIGIBILITY:
Inclusion:

1. Penn State Worry Questionnaire (trait) score meeting threshold of 65 or higher.
2. Endorsement of symptoms consistent with Generalized Anxiety Disorder on the MINI interview with a CSR equal to or greater than 4.
3. If other symptoms are present, associated CSR is at least 1 point lower than the CSR associated with GAD symptoms

Exclusion

1. Having a current or past history of mania or psychosis, or endorsement of symptoms consistent with a substance use disorder in the past 12 months.
2. Reporting of suicidal ideation, intent or plan.
3. Participants are excluded if they are currently receiving psychological treatment or counseling unless this treatment is infrequent (meeting once monthly or less) or the participant has been receiving consistent weekly treatment for 12 weeks and still meets all other eligibility criteria.
4. Psychotropic medication with a change in dose in the past 12 weeks. If they have recently discontinued a psychotropic medication, they will be included if it has been at least 1 month since discontinuation or 3 months in the case of fluoxetine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2015-06-12 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2019-10-28 (Actual)

PRIMARY OUTCOMES:
Change in worry as measured by the Penn State Worry Questionnaire - Past Week | this measure is administered at baseline, at post-test (1 week post baseline), at 1 week follow up and at 1 month follow up

SECONDARY OUTCOMES:
Change in depressive symptoms as measured by the Centre for Epidemiological Studies Depression Scale | this measure is administered at baseline, at post-test (1 week post baseline), at 1 week follow up and at 1 month follow up
Change in negative problem orientation as measured by the Negative Problem Orientation Questionnaire | this measure is administered at baseline, at post-test (1 week post baseline), at 1 week follow up and at 1 month follow up
Change in quality of problem-solving as measured by The Means-Ends Problem-Solving task | this measure is administered at baseline, at post-test (1 week post baseline), at 1 week follow up and at 1 month follow up
Change in problem solving style as measured by the Social Problem Solving Inventory Revised | Administered at baseline, at post-test (1 week post baseline), at 1-week follow up and at 1-month follow up
Change in attentional control as measured by the Attentional Control Scale | this measure is administered at baseline, at post-test (1 week post baseline), at 1 week follow up and at 1 month follow up
Change in residual working memory capacity as measured by the Random Interval Generation Task | this measure is administered at baseline, at post-test (1 week post baseline), at 1 week follow up and at 1 month follow up
- Change in interpretation bias as measured by the Ambiguous/ Unambiguous Situations Diary Extended | this measure is administered at baseline, at post-test (1 week post baseline), at 1 week follow up and at 1 month follow up
Change in cognitive avoidance as measured by the Cognitive Avoidance Questionnaire | this measure is administered at baseline, at post-test (1 week post baseline), at 1 week follow up and at 1 month follow up
Change in worry as measured by experience sampling completed during the 7 days between baseline and post test | Daily during 7-day intervention period
Change in affect as measured by experience sampling completed during the 7 days between baseline and post test | Daily during 7-day intervention period
Change in concreteness as measured by experience sampling completed during the 7 days between baseline and post test. | Daily during 7-day intervention period
Change in GAD-Q-IV severity | this measure is administered at baseline, at post-test (1 week post baseline), at 1 week follow up and at 1 month follow up

OTHER OUTCOMES:
Change in trait anxiety as measured by STICSA | Administered at baseline, at post-test (1 week post baseline), at 1-week follow up and at 1 month follow up
Change in mood/affect as measured by PANAS | Administered at baseline, at post-test (1 week post baseline), at 1-week follow up and at 1-month follow up.
Change in intolerance of uncertainty as measured by the Intolerance of Uncertainty Scale | Administered at baseline, at post-test (1 week post baseline), at 1-week follow up and at 1-month follow up
Change in emotion dysregulation as measured by the DERS | Administered at baseline, at post-test (1 week post baseline), at 1-week follow up and at 1-month follow up
Change in distress tolerance as measured by the Distress Tolerance Scale | Administered at baseline, at post-test (1 week post baseline), at 1-week follow up and at 1-month follow up
Change in imagery use as measured by the Spontaneous Use of Imagery Scale [ | Administered at baseline, at post-test (1 week post baseline), at 1-week follow up and at 1-month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Koerner, PhD, Principal Investigator — Toronto Metropolitan University
Locations (1):
- Psychology Research and Training Centre, Ryerson University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Watkins ER, Baeyens CB, Read R. Concreteness training reduces dysphoria: proof-of-principle for repeated cognitive bias modification in depression. J Abnorm Psychol. 2009 Feb;118(1):55-64. doi: 10.1037/a0013642. PMID 19222314
- [Background] Borkovec TD, Inz J. The nature of worry in generalized anxiety disorder: a predominance of thought activity. Behav Res Ther. 1990;28(2):153-8. doi: 10.1016/0005-7967(90)90027-g. PMID 2183759
- [Background] Stöber, J. & Borkovec, T.D. (2002). Reduced concreteness of worry in generalized anxiety disorder: Findings from a therapy study. Cognitive Therapy and Research, 26, 89 - 95.